CLINICAL TRIAL: NCT04002011
Title: Oral Anticoagulation After Cardiac Surgery in the Era of Direct Oral Anticoagulants: is Large Use of Vitamin K Antagonists Still Justified?
Brief Title: DOAC Versus VKA After Cardiac Surgery
Acronym: DOAC/VKA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Submission process abandoned. No patient enrolled.
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Pierre Voisine, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21755
Record Dates: First submitted 2019-06-10; First posted 2019-06-28 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Anticoagulant-induced Bleeding
Keywords: direct oral anticoagulant; vitamin K antagonist; cardiac surgery; perioperative care
MeSH Terms: interventions — Warfarin; Dabigatran; Rivaroxaban; apixaban; edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group VKA (Active Comparator): 103 patients. First intake at postoperative day 1 or later when anticoagulation is secondary indicated.
  Dosage adapted to INR = [2.0-3.0], parenteral (subcoutaneous low-weight molecular or intravenous unfractionated heparin) until INR > or = 2.0.
  Daily INR during hospital stay, then management by familial doctor. Duration: 3 months
  Interventions: Drug: Warfarin
- Group DOAC (Active Comparator): 103 patients - One drug among the 4 DOAC according the morbidity of each patient (preoperative DOAC, oral nutrition recovery).
  First intake at hospital discharge - parenteral (subcoutaneous low-weight molecular or intravenous unfractionated heparin) during hospital stay.
  Regular daily dosages according the drug, its indication (atrial fibrillation/flutter or biological mitral replacement/repair or biological tricuspid replacement versus venous thromboembolism) and the morbidity of each patient (age, weight, creatinine ou its clearance).
  Validation by one referent pharmacist. No biological monitoring. Duration: 3 months
  Interventions: Drug: Dabigatran; Drug: Rivaroxaban; Drug: Apixaban; Drug: Edoxaban

INTERVENTIONS:
Drug: Warfarin — It will be started on postoperative day 1 or later when oral anticoagulation is secondary indicated. Daily dose will be adapted to obtain an international normalized ratio of [2.0-3.0]. Other anticoagulants will be not administrated.
  Other Names: Coumadin
  Arms: Group VKA
Drug: Dabigatran — It will be started when patients will be discharged from our center. Our pharmacist referent will validated the drug and its daily dose. Other anticoagulants will be not administrated.
  Other Names: Pradaxa
  Arms: Group DOAC
Drug: Rivaroxaban — It will be started when patients will be discharged from our center. Our pharmacist referent will validated the drug and its daily dose. Other anticoagulants will be not administrated.
  Other Names: Xarelto
  Arms: Group DOAC
Drug: Apixaban — It will be started when patients will be discharged from our center. Our pharmacist referent will validated the drug and its daily dose. Other anticoagulants will be not administrated.
  Other Names: Eliquis
  Arms: Group DOAC
Drug: Edoxaban — It will be started when patients will be discharged from our center. Our pharmacist referent will validated the drug and its daily dose. Other anticoagulants will be not administrated.
  Other Names: Lixiana
  Arms: Group DOAC

SUMMARY:
Postoperative management of oral anticoagulation is a frequent preoccupation in cardiac surgery, concerning about half of patients. Vitamin K antagonists are often recommended but their management is not easy due to the high dose-response patient variability. Pharmacologically more stable, direct oral anticoagulants have similar efficiency in preventing thromboembolic complications while they decrease the risk of bleeding in certain patient populations. The objective of study is to assess the safety and efficacy of direct oral anticoagulants in the postoperative period of cardiac surgical procedures.

DETAILED DESCRIPTION:
This study will be composed by 2 groups of 103 participants, patients undergoing cardiac surgery and needing oral anticoagulation in the early postoperative period.

The control group will receive vitamin K antagonist and the study group will receive direct oral anticoagulant. The investigators will call back each participants at 3 months to report the ischemic and bleeding complications during this period and evaluated the quality of life of the oral anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery, with or without cardiopulmonary bypass
* Indication of postoperative oral anticoagulation: preoperative (atrial fibrillation/flutter of idiopathic venous thromboembolism disease), intraoperative (bioprosthetic mitral valve replacement/mitral valve repair or bioprosthetic tricuspid valve repair), postoperative (de novo persistent more than 24 hours or recurrent atrial fibrillation/flutter, venous thromboembolism)

Exclusion Criteria:

* mechanical valvular prostheses or ventricular assist devices
* morbidly obesity (body mass index ≥ 40 kg/m²), prior biliopancreatic diversion or sleeve gastrectomy
* perioperative dysphagia needing naso-enteric tube or jejunostomy
* antiretroviral of antifungal oral therapy
* perioperative recent (less than 2 weeks) stroke
* perioperative severe renal failure (clearance of creatinine under 30 mL/min or dialysis)
* perioperative severe hepatic failure (elevated alanine aminotransferase more than 3 times the superior limit of normal range or cirrhosis)
* perioperative recent (less than 3 months) heparin-induced thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-09 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Hemorrhagic events with anticoagulant treatment | Evaluation at month 3 after hospital discharge for all the postoperative period
  The investigators will use the regional computerized medical record of each participants to report all the hemorrhagic event during all the postoperative period, and define them according the "Bleeding Academic Research Consortium" (BARC) criteria. Hemorrhage-free survival will be studied.
Ischemic events with anticoagulant treatment | Evaluation at month 3 after hospital discharge for all the postoperative period
  The investigators will use the regional computerized medical record of each patients to report all the ischemic event during all the postoperative period. Ischemia-free survival will be studied.
Death with anticoagulant treatment | Evaluation at month 3 after hospital discharge for all the postoperative period
  The investigators will use the regional computerized medical record of each patients to report all the ischemic event during all the postoperative period. Global survival will be studied. Ischemic or hemorrhagic death will be precised.
Quality of life with anticoagulant treatment | Evaluation at month 3 after hospital discharge for the last month
  The investigators will call back all the participants by phone and use the SF-12 questionnaire (score between 12 and 56) to evaluate the quality of life about several dimensions (global, physic, mental, pain, society).
Statisfaction of the anticoagulant treatment | Evaluation at month 3 after hospital discharge for the last month
  The investigators will call back all the participants by phone and use the anti-clot treatment scale (ACTS) to evaluate the feelings of "burdens" (score between 12-60) and "benefits" (score between 3-15) of the anticoagulant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Voisine, M.D., Principal Investigator — Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ)